CLINICAL TRIAL: NCT04006626
Title: 18F-FES PET/CT Influences the Staging and Management of Newly Diagnosed Oestrogen Receptor-Positive Breast Cancer Patients: A Retrospective Comparative Study With 18F-FDG PET/CT
Brief Title: 18F-FES PET/CT's Additional Clinical Value in ER+ BC
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-7
Record Dates: First submitted 2019-06-26; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PET group: the staging and management of newly diagnosed ER+ Breast Cancer Patients based on 18F-FDG PET/CT
- FES group: the staging and management of newly diagnosed ER+ Breast Cancer Patients based on 18F-FDG PET/CT and 18F-FES PET/CT

SUMMARY:
To figure out whethetr 18F-FES PET/CT could influence the staging and management of newly diagnosed Oestrogen Receptor-positive Breast Cancer Patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed immunohistochemical confirmed oestrogen receptor (ER)-positive breast cancer
* Patients underwent both 18F-FES PET/CT and 18F-FDG PET/CT in Fudan University Shanghai Cancer Center within 1 week after diagnosis
* Patients with available medical history

Exclusion Criteria:

* Patients with incomplete medical history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Staging of breast cancer | 6 weeks
  Deliver questionnaire to phycians to investigate the staging of BC according to AJCC 8 (TNM staging).

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Biyun Wang, MD, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided